Title: A feasibility pilot study for a social support intervention in kidney transplant candidates

NCT Number: NCT04363515

Date: October 1, 2024

## Statistical analysis plan

As outlined in protocol section 6.3, this is a feasibility pilot study; therefore, it is not powered to test anything. We will be collecting data that we could adjust for (i.e. demographics), but we will not be adjusting, because the main goal of this particular study is to gauge if the intervention is feasible.